CLINICAL TRIAL: NCT00322712
Title: INST 0603C Chart Review on Patients With Unresectable/Metastatic Pancreatic Cancer Treated in the UNM Cancer
Brief Title: INST 0603C Patients With Unresectable/Metastatic Pancreatic Cancer Treated in the UNM Cancer
Status: Terminated | Type: Observational
Why Stopped: This is only a chart review. This is not a clinical trial and was inadvertently entered in the system.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: INST 0603C
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Chart Review of patients with pancreatic cancer treated with combination of irinotecan, oxaliplatin and cetuximab.

DETAILED DESCRIPTION:
Chart Review to describe the clinical outcomes in patients pancreatic cancer treated with combination of irinotecan, oxaliplatin and cetuximab.

ELIGIBILITY:
Inclusion Criteria:

Patients with unresectable/metastatic pancreatic cancer treated in the UNM Cancer Research and Treatment Center.

Exclusion Criteria:

Not specified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable/metastatic pancreatic cancer treated in the UNM Cancer Research and Treatment Center.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fa-Chyi Lee, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Retrospective chart review for the period from 10/2005-8/2006 done on all patients with metastatic pancreatic cancer treated at the UNM Cancer Center with OIC (Oxaliplatin 60mg/m2, Irinotecan 90mg/m2, and Cetuximab 250 mg/m2 delivered every other week).
Period: Overall Study
Arm/Group | Treatment Arm
Started | 12
Completed | 11
Not Completed | 1
Not completed — treated with bevacizumab not cetuximab | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: Years] | 70 [50 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Time to Death
Description: Length of survival of patients treated with a combination of Oxaliplatin 60mg/m2, Irinotecan 90mg/m2, and Cetuximab 250 mg/m2 delivered every other week.
Time Frame: From date of treatment until time of death
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
Months | 7 [3 to 18]

ADVERSE EVENTS:
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes